CLINICAL TRIAL: NCT00827788
Title: The Contrast Media and Nephrotoxicity Following Coronary Revascularization by Primary Angioplasty for Acute Myocardial Infarction. The CONTRAST-AMI Study.
Brief Title: Comparison Between Iso-Osmolar and Ipo-Osmolar Contrast Agents in Patients With Acute Myocardial Infarction (AMI) Undergoing Primary Percutaneous Coronary Intervention (PCI)
Acronym: CONTRAST-AMI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ospedale San Donato (Other)
Collaborators: Ospedale Le Scotte (Other); Ospedale della Misericordia - Grosseto (Unknown)
Responsible Party: Cardiovascular Department USL 8(Leonardo Bolognese MD), Ospedale SanDonato
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Arezzo001; EUDRACT 2008-008491-13
Record Dates: First submitted 2009-01-22; First posted 2009-01-23 (Estimated); Last update posted 2010-11-16 (Estimated); Status verified 2009-09

CONDITIONS: Contrast Induced Nephropathy; Acute Myocardial Infarction
Keywords: contrast media; angiography; percutaneous coronary intervention
MeSH Terms: interventions — iodixanol; iopromide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- iodixanol (Active Comparator): Iso-osmolar contrast medium (Iodixanol) will be administered during PCI
  Interventions: Drug: Iodixanol
- iopromide (Active Comparator): Low-osmolar contrast medium (Iopromide) will be administered during PCI
  Interventions: Drug: Iopromide

INTERVENTIONS:
Drug: Iodixanol — Iso-osmolar contrast medium (Iodixanol) will be administered during PCI
  Other Names: Visipaque®
  Arms: iodixanol
Drug: Iopromide — Low-osmolar contrast medium (Iopromide) will be administered during PCI
  Other Names: Ultravist®
  Arms: iopromide

SUMMARY:
The purpose of this study is to determine the incidence of contrast induced nephropathy and myocardial tissue reperfusion following iso-osmolar iodixanol or ipo-osmolar iopromide administration in patients with acute myocardial infarction undergoing primary PCI.

DETAILED DESCRIPTION:
This is a multicentric randomized comparison between iso-osmolar and ipo-osmolar contrast agents in patients treated with primary PCI with the evaluation of contrast-induced nephropathy incidence and myocardial tissue reperfusion. The study was designed as a non-inferiority trial.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged ≥ 18
* Patients with ST-elevation Myocardial Infarction presenting within 12 hours after the onset of symptoms (18 hours in case of cardiogenic shock), who are scheduled to undergo primary PCI
* Patients who have signed and dated the written informed consent form

Exclusion Criteria:

* Patients in pregnancy or lactation
* Long-term dialysis
* Administration of any investigational drug within the previous 30 days
* Intra-arterial or intravenous administration of iodinated contrast medium from 7 days before to 72 hours after the administration of study drug
* Intake of any nephrotoxic medications 24 hours before or after the administration of study drug
* Contraindications to the study drug or the cardiac catheterization procedure
* Previous participation in this study
* As the discretion of the investigator, the patient has any conditions not appropriate to the usage of iodinated contrast agent or not appropriate to undergo cardiac catheterization procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 432 (Estimated)
Dates: Start 2008-12; Primary Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Incidence of Contrast Induced Nephropathy (CIN) between the two study groups, defined as relative increase of serum Creatinine of 25% or more from basal values | days 1, 2, 3, and at discharge

SECONDARY OUTCOMES:
TIMI grade flow | before and after primary PCI
Corrected TFC (TIMI frame count) | after primary PCI
TMPG (TIMI Myocardial Perfusion Grade) | after PCI
LFR slope (load to function slope) | after primary PCI
MACE | 1, 6, 12 months
absolute increase in serum Creatinine | days 1, 2, 3, and at discharge
relative increase in serum creatinine of 50% or more | days 1, 2, 3, and at discharge

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo Bolognese, MD, FESC, Principal Investigator — Ospedale SanDonato
Locations (1):
- Cardiovascular Department, Ospedale S.Donato, Arezzo, AR, Italy

REFERENCES:
- [Derived] Bolognese L, Falsini G, Grotti S, Limbruno U, Liistro F, Carrera A, Angioli P, Picchi A, Ducci K, Pierli C. The contrast media and nephrotoxicity following coronary revascularization by primary angioplasty for acute myocardial infarction study: design and rationale of the CONTRAST-AMI study. J Cardiovasc Med (Hagerstown). 2010 Mar;11(3):199-206. doi: 10.2459/JCM.0b013e32833186a4. PMID 19829124